CLINICAL TRIAL: NCT04296110
Title: Impact of a Biofeedback Intervention on Microbiome, Metabolome, and Clinical Outcomes in Pediatric IBD(Study 2).
Brief Title: Impact of a Biofeedback Intervention on Microbiome, Metabolome, and Clinical Outcomes in Pediatric IBD (Study 2)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues with study funding
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Ross Maltz, Principal Investigator, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01100
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: IBD
Keywords: biofeedback; pediatric
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants will receive music relaxation therapy. They will be asked to listen to designated music daily for 12 weeks.
  Interventions: Other: Music Relaxation Therapy
- Biofeedback (Experimental): Participants will receive a biofeedback intervention. They will be asked to practice breathing at their designated resonance frequency using provided biofeedback device daily for 12 weeks.
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Behavioral: Biofeedback — They will also be taught how to use the biofeedback app and Inner Balance device. Additionally, they will also be educated on the principles of biofeedback and its benefits and taught how to maximize HRV by using self-regulation breathing techniques.They will be given an Inner Balance device, which is an ear sensor that connects to an apple device that measures heart rate variability (HRV) and gives them access to an app that is designed to help them improve their HRV. They will be asked to practice breathing at their resonance frequency using the Inner Balance device daily for 5-15 mins for the duration of the 12-week intervention. Patients and the research coordinator will have access to all of their sessions and results. The research coordinator will monitor compliance via the Heartcloud associated with their device and encourage adherence throughout the intervention.
  Other Names: Inner Balance
  Arms: Biofeedback
Other: Music Relaxation Therapy — We will determine what genre of music is most relaxing to them and ask them to listen to this type of music using the spotify app for 5-15 mins a day for 12 weeks. If they do not have access to a device that they can listen to spotify on, an ipod will be provided. They will be asked to complete a 2-question survey via Redcap daily that asks them if they have listened to the designated music that day and for how long.
  Other Names: MRT
  Arms: Control

SUMMARY:
This prospective, randomized, longitudinal, controlled study will enroll pediatric CD patients with inflammatory, non-stricturing, and non-penetrating disease type with mild/quiescent disease based on Pediatric Crohn's Disease Activity Index (PCDAI). Participants will be randomized to receive HRV biofeedback intervention daily for 12 weeks or to music relaxation therapy.

DETAILED DESCRIPTION:
The inflammatory bowel diseases (IBD), which include Crohn's disease (CD) and ulcerative colitis (UC), affects 3 million Americans. In approximately 25-30% of patients, onset of these chronic diseases occurs prior to the age of 20. Despite medical advances in new therapies, the clinical remission rate on biologics is less than 50% and a significant number of patients will lose response to anti-TNF therapy over time. In addition, patients that require a change in therapy will have a lower response rate to a different biologic. Additional therapies and mechanisms that affect disease activity need to be investigated to identify complimentary treatments that can further impact remission rates without increasing side effects such as lymphoma.

Environmental factors, such as stressor exposure, can exacerbate mucosal inflammation. Patients with IBD report a lower quality of life, as well as increased anxiety and depression. Psychological interventions may improve disease activity. This study will test, using a randomized clinical trial (RCT) design, whether biofeedback intervention will attenuate disease activity. If efficacious, this study will provide a rationale for establishing biofeedback as a complimentary therapy to standard of care to ameliorate stress-induced increases in chronic inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-17 years
2. Have inflammatory, non-stricturing, and non-penetrating CD with either mild/quiescent disease based on PCDAI or PGA
3. Live within a 2 hour drive of NCH

Exclusion Criteria:

1. Participants are excluded if they have ulcerative colitis, penetrating and/or stricturing CD, have a comorbid chronic illness, perianal disease, taking antibiotics within the last 3 months, psychological disorders that they are undergoing treatment or taking medication for at that time, presence of a heart rhythm or other abnormality of heart rhythm on screening EKG, or undergoing psychological treatments such as cognitive behavioral therapy, mindfulness, or biofeedback therapy at the time of enrollment.
2. Age and language are limited by the demands of the study (questionnaire completion

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Disease activity( Fecal calprotectin) | enrollment to 12 month follow up
  Fecal calprotectin levels from stool
Disease Activity (Crohn's disease) | enrollment to 12 month follow up
  Pediatric Crohn's Disease Activity Index total score. A standard measure of disease severity that is comprised of information obtained from patient recall (pain severity, stool frequency, limitation of activities), examination (weight, height, abdominal tenderness, perirectal disease, extra- intestinal manifestations), and laboratory data. The Pediatric Crohn's Disease Activity Index total score will be used from baseline, post-intervention, 3 months post-intervention, and 12 month follow up. Higher scores indicate more severe disease. Scores range from 0-100.
Stress | enrollment to 12 month follow up
  PROMIS Pediatric Psychological Stress Experiences.Scores range from 0-60, with higher scores indicating higher levels of stress.Total score will be used from baseline, post-intervention, 3 months post-intervention, and 12 month follow up.
Anxiety | enrollment to 12 month follow up
  PROMIS Pediatric Anxiety Short Form. Scores range from 0-60, with higher scores indicating higher levels of anxiety. Total score will be used from baseline, post-intervention, 3 months post-intervention, and 12 month follow up.
Pediatric Quality of Life: scale | enrollment to 12 month follow up
  PedsQL. Scores range from 0-100 with higher scores indicating higher quality of life. Total score will be used from baseline, post-intervention, 3 months post-intervention, and 12 month follow up.
Depression | enrollment to 12 month follow up
  Children's Depression Inventory short form. Scores range from 0-54, with higher scores indicating higher levels of depression. Total score will be used from baseline, post-intervention, 3 months post-intervention, and 12 month follow up.

SECONDARY OUTCOMES:
Stress-related changes in the microbiome | enrollment to 12 month follow up
  Microbiome α and β-diversity will be examined at baseline, post-intervention, 3 month post-intervention, and 12 month follow-up to determine possible relationships between overall community structure between participants that received the intervention of biofeedback vs participants that were controls.
Stress-related changes in the metabolome. | enrollment to 12 month follow up
  Random Forest (RF) and Boruta feature selection will be used from baseline, post-intervention, 3 month post-intervention, and 12 month follow-up to identify metabolites and microbes.To further interpret the biological function of predictive metabolites, pathway enrichment analysis will be performed using the RaMP database, which integrates biological pathway and metabolite annotions from multiple sources (e.g. HMDB, KEGG, REACTOME, WikiPathways).

CONTACTS AND LOCATIONS:
Overall Officials: Ross Maltz, MD, Principal Investigator — Nationwide Childrens Hospital
Locations (1):
- Nationwide Childrens Hospital GI Clinic, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No